CLINICAL TRIAL: NCT05303480
Title: An Exploratory, Single-centre, Two-part Study to Describe Mycosis Fungoides Characteristics and Explore Novel Biomarkers With a Multi- Modal Patient Profiling Approach by Comparing MF Patients to Healthy Volunteers
Brief Title: Deep Phenotyping of Cutaneous T Cell Lymphoma, Type Mycosis Fungoides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Human Drug Research, Netherlands (Other)
Collaborators: RECORDATI GROUP (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHDR1947; 2021-001576-41 (EudraCT Number); NL77292.056.21 (Other: Regulatory registration number)
Record Dates: First submitted 2021-12-07; First posted 2022-03-31 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-03

CONDITIONS: Mycosis Fungoides
Keywords: Mycosis Fungoides; Cutaneous T Cell Lymphoma; Biomarker; Chlormethine; Ledaga
MeSH Terms: conditions — Mycosis Fungoides; Lymphoma, T-Cell, Cutaneous | interventions — Mechlorethamine; Amines

STUDY DESIGN:
Intervention Model Description: This is an observational and interventional study in 20 Mycosis Fungoides patients and 10 healthy volunteers (observational only).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chlormethine gel (Active Comparator): Chlormethine gel 0.016% in 60mg tube, topical home administration from day 0 to day 155.
  Interventions: Drug: Chlormethine
- Healthy volunteers (No Intervention): Healthy volunteer cohort (observational)

INTERVENTIONS:
Drug: Chlormethine — Chlormethine gel 0.016%
  Other Names: Ledaga; Valchlor
  Arms: Chlormethine gel

SUMMARY:
Mycosis fungoides (MF) is an ultra-orphan disease of which the etiology remains unknown. MF is diagnosed by correlating clinical appearance with histopathological analysis of often multiple invasive skin punch biopsies. To move patient care and the development of novel treatments for MF forward, objective, sensitive and reliable tools that are preferably non-invasive are desired. Therefore, the objective of the current study is to phenotype the early stages of mycosis fungoides in detail and to assess the response of chlormethine (CL) gel monotherapy. With this approach the investigators aim to detect novel biomarkers and to establish methodologies for the (non-)invasive monitoring of MF.

DETAILED DESCRIPTION:
In recent years, knowledge about the wide spectrum of cutaneous T-cell lymphomas (CTCL) has broadened. Mycosis fungoides (MF) comprises about 50-70% of all primary cutaneous T-cell lymphomas (Willemze et al, 2019). Many CTCL are misdiagnosed due to clinical and histopathological similarity to other skin conditions (such as psoriasis vulgaris, atopic dermatitis and tinea corpora), low prevalence of disease and a lack of reliable tools for detection of these diseases, resulting in delayed diagnosis with years of discomfort and possibly a worse prognosis. Furthermore, standard treatment has never been proven curative, has many side effects and exacerbations are frequent. To date, the etiology of mycosis fungoides remains unknown and little research has been conducted into the mechanisms underlying its development and its response to treatment.

Mycosis fungoides lesions change over time and differ between patients, consisting of three morphologically different stages: patches (erythematosquamous maculae), plaques (erythematosquamous, elevated and occasionally infiltrated lesions) and tumors (with or without ulceration). Only a relatively small group of patients advances to tumor stage MF during their lifetime. Mycosis fungoides is diagnosed by correlating clinical appearance with histopathological analysis of an invasive skin punch biopsy. Additionally, often multiple biopsies are required after diagnosis, e.g. when a lesion is clinically advancing to a different stage or if lesion origin is ambiguous. Currently no other biomarkers besides skin punch biopsies markers are available for the diagnosis of MF, the evaluation of a MF lesion over time, and the monitoring of a potential treatment effect. To advance MF patient care and the development of novel treatments for MF objective, sensitive and reliable (preferably non-invasive) tools are desired.

Therefore, the objective of the current study is to evaluate disease-related characteristics and biomarkers, the intra- and inter-patient variability of biomarkers, to evaluate biomarkers for disease-monitoring following CL gel treatment and to investigate and monitor skin-related adverse events that might develop after CL gel application in MF patients. With this approach the investigators aim to detect novel biomarkers and to establish methodologies for the (non-)invasive monitoring of MF.

For this purpose, a multi-modal patient profiling approach with in-depth characterization of cutaneous T-cell lymphomas will be performed. A clinical study will be conducted investigating the biology of the disease compared to healthy volunteers (part A) and patients' response to intervention (part B). The former to characterize objectively measured disease characteristics and mechanisms underlying its development, the latter to monitor the biomarker response associated to a MF-CTCL treatment, in this case CL gel. The study focusses on cellular, molecular, biophysical, imaging and microbiome analyses in comparison to healthy controls and between lesional and non-lesional skin of MF patients.

ELIGIBILITY:
Healthy volunteers must meet all of the following inclusion criteria:

1. Signed informed consent prior to any study-mandated procedure;
2. Male or female subjects, 18 to 75 years of age, inclusive at screening; in general, stable good health as per judgement of the investigator based upon the results of a medical history, physical examination, vital signs, ECG and laboratory assessments performed at screening. Repeated laboratory testing may be performed at the discretion of the clinical investigators;
3. Body mass index (BMI) ≥ 18.0 and ≤ 40.0 kg/m2; during COVID-19 pandemic only ≥ 18.0 and ≤ 33.0 kg/m2;
4. No clinically significant skin disease as judged by the investigator;
5. No history of hypertrophic scarring or keloid;
6. Subject is willing to refrain from extensively washing (including bathing, swimming, showering and excessive sweating) the skin 4 hours before every study visit;
7. Subject is willing and able to washout and withhold any topical treatment (prescription and over the counter products) in the treatment area (if possible matched location to most common location of target lesions of the MF group, and otherwise 100cm2 on the lower back) for 2 weeks prior to Day 1;
8. Subject is willing to refrain from application of any topical product (e.g. ointments, crème or washing lotions) on the skin 24 hours prior to every study visit day;
9. Subject is willing and able to washout (topical and oral) antibiotic therapy for 14 days prior to Day 1;
10. Subject is willing to use effective contraception from screening until EOS if subject is male or women of childbearing potential;
11. Subject has the ability to communicate well with the investigator in the Dutch language and is willing to comply with the study requirements.

Eligible MF patients must meet all of the following inclusion criteria at screening:

1. Signed informed consent prior to any study-mandated procedure;
2. Male or female subjects, 18 to 75 years of age, inclusive at screening; in general, stable good health as per judgement of the investigator based upon the results of a medical history, physical examination, vital signs, ECG and laboratory assessments performed at screening. Repeated laboratory testing may be performed at the discretion of the clinical investigators
3. Body mass index (BMI) ≥ 18.0 and ≤ 40.0 kg/m2; during COVID-19 pandemic only ≥ 18.0 and ≤ 33.0 kg/m2;
4. At least one patch and/or plaque lesion present, with at least one dimension with a diameter of ≥ 6cm;
5. Confirmed MF-diagnosis (stage 1a/1b) by histology (or clinico-histopathological correlation) within the last 10 years;
6. Willing and able to washout any topical treatment for MF (at least 2 weeks) and any systemic treatment for MF (at least 4 weeks) prior to Day 1, resulting in a washout of 8 weeks for topical treatment and 10 weeks for disease-related systemic treatment prior to the first dosing day (day 43);
7. No previous use of CL gel (Ledaga) in the past two years;
8. Subject is willing and able to washout (topical and oral) antibiotic therapy for 14 days prior to Day 1;
9. Subject is willing to refrain from extensively washing (including bathing, swimming, showering and excessive sweating) the skin 6 hours before every study visit day and up to 2 hours after application of the treatment gel;
10. Subject is willing to use effective contraception during the study if subject is male or women of child bearing potential, for up to 90 days after the last dose of study treatment;
11. Male subjects must be willing to withhold from any sperm donation during the study and up to 90 days after the last dose of study treatment.

Eligible healthy volunteers must meet none of the following exclusion criteria at screening:

1. History of immunological abnormality (e.g., immune suppression) that may interfere with study objectives, in the opinion of the investigator;
2. The use of systemic antibiotic therapy for >2 months the past 12 months;
3. The use of any oral/systemic medication (e.g. immunomodulatory, immunosuppressive) within 28 days prior to Day 1, if the investigator judges that it may interfere with the study objectives.
4. Positive hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV ab), or human immunodeficiency virus antibody (HIV ab) at screening;
5. Participation in an investigational drug study within 3 months prior to screening or more than 4 times a year;
6. Loss or donation of blood over 500mL within three months prior to screening;
7. History of alcohol consumption exceeding 5 standard drinks per day on average within 3 months of screening. Alcohol consumption will be prohibited from at least 24 hours preceding each study visit;
8. Positive urine test for drugs or history of abuse at screening or pre-dose. Urine drug test may be repeated at the discretion of the investigator;
9. Pregnant, a positive pregnancy test, intending to become pregnant, or breastfeeding;
10. Any other known factor, condition, or disease that might interfere with study conduct or interpretation.

    Eligible MF-patients must meet none of the abovementioned and following exclusion criteria at screening:
11. Have any current relevant skin infections/disease in the treatment area other than the observational disease (mycosis fungoides), inclusively, but not limited to atopic dermatitis, psoriasis vulgaris, dermatomycosis and other skin malignancies.
12. Having received treatments for MF or any other disease within the following intervals prior to the start of the study (The use of topical emollients is allowed during the study. For target lesions it is allowed up to 24h before every study visit day):

    1. < 2 weeks for topical treatment, e.g. corticosteroids, retinoids, vitamin D analogs
    2. <4 weeks for phototherapy, e.g. UVB, PUVA, PDT
    3. <4 weeks for non-biologic systemic treatment, e.g. retinoids, methotrexate
    4. <6 weeks for peginterferon alfa-2a
    5. <8 weeks for radiotherapy or surgery in the treatment area
    6. <3 months for any systemic chemotherapeutical treatment
13. Known hypersensitivity to chlormethine gel or its excipients.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

PRIMARY OUTCOMES:
Composite Assessment of Index Lesions Disease Severity Score (CAILS) | from day -42 to day 155
  CAILS is a composite score to quantify lesion severity and consists of scoring erythema, hypo-/hyperpigmentation, plaque elevation, desquamation and lesion size. The CAILS score of a single lesion ranges from 0 (unaffected) to 50 (severely affected).
Modified Severity Weighted Assessment Tool (mSWAT) | from day -42 to day 155
  mSWAT combines the assessment of the severity of lesions and the area affected into a single score ranging from 0 (unaffected) to 400 (severely affected).
Objective Response Rate (ORR) | from day 43 to day 155
  The Objective Response Rate (ORR) measures the lesional response as the change from baseline for the CAILS and mSWAT score. The ORR is the number of patients with complete response (100% clearance) + the number of patients with partial response (50%-99%) divided by the total number of patients.
SKINDEX-29: Quality of life (QoL) | from day 0 to day 155
  The Skindex-29 is a valid 29-item self-report measure that evaluates health-related QoL for patients with dermatological diseases. The score is subdivided in a domain for symptoms, emotions and fuctioning; domain scores range from 0 (no impact) to 100 (severely impacted). Total Skindex-29 score is calculated as a mean of the three domains, ranging from 0 (no impact on QoL) to 100 (QoL severely impacted).
Treatment Satisfaction Questionnaire for Medication (TSQM) | from day 43 to day 155
  TSQM consists of 14 questions and explores the subject satisfaction regarding the effectiveness, the side effects, convenience and global satisfaction of the investigational drug. The TSQM score ranges from 0 (lowest satisfaction) to 100 (highest satisfaction).
Patient reported outcomes | from day 0 to day 155
  Patients will be asked to report on their condition through a Numerical Rating Scale (0 (better)- 100 (worse)) for itch, pain and sleeplessness.
Erythema measurement of the skin | from day 0 to day 155
  Redness of the skin will be determined using a colorimeter
3D Multispectral imaging | from day 0 to day 155
  The redness and superficial morphology of (non-)lesional skin sites will be determined using a 3D multispectral imaging system.
Laser Speckle Contrast Imaging (LSCI) | from day 0 to day 155
  The cutaneous microcirculation of (non-)lesional skin sites will be monitored over a 40 second timespan with a laser speckle contrast imager.
Thermography | from day 0 to day 155
  Body surface temperature of (non-)lesional skin will be determined using a thermal imaging infrared camera.
Optical Coherence Tomography (OCT) | from day 0 to day 155
  OCT is a non-invasive assessment which visualizes skin morphology in vivo to a depth of 2 mm with the use of infrared light.
Skin barrier function by Trans-Epidermal Water Loss (TEWL) | from day 0 to day 155
  The barrier status by trans epidermal water loss of (non-)lesional skin will be determined using TEWL. (g/m2/h)
Cutaneous microbiome | from day 0 to day 155
  The cutaneous microbiome of (non-)lesional skin is collected by swabbing. The abundance of bacteria is thereafter determined using next-generation sequencing.
Faecal microbiome | from day 43 to day 155
  The bacterial composition of stool samples pre- and post-treatment will be determined using next-generation sequencing.
Skin surface biomarkers | from day 0 to day 155
  Superficial protein biomarkers of (non-)lesional skin will be assessed by a non-invasive transdermal patch by FibroTx. The presence of protein biomarkers will be determined using ELISA.
  The following biomarkers will be assessed (ng/ul): IL-8, CXCL-2, IL-1A, IL-1RA, CCL-17 and CCL-27 and VEGF.
Lipidomics of the stratum corneum by liquid chromatography mass spectroscopy | from day 0 to day 155
  Tape stripping will be performed on (non-)lesional skin and lipids are subsequently extracted from the tape and analyzed using Liquid Chromatography-Mass Spectrometry (ng/cm2).
Patient genotyping | day 43
  A whole blood sample will be used to scan for common mutations in genes implicated in mycosis fungoides using next-generation sequencing.
Blister immune cell subsets | day 43
  Blisters will be induced on the (non-)lesional skin and the blister exudate aspirated. Blister exudate will be analyzed for the presence of immune cells (e.g. CD4+ and CD8+ T-Cells) using flow cytometry.
Blister protein biomarkers by high-throughput, multiplex immunoassays of proteins by Proximity Estension Assay (PEA) technology | day 43
  Blisters will be induced on the (non-)lesional skin and blister fluid aspirated. Blister fluid will be analyzed for the presence of various chemokines and cytokines using the Olink inflammation and immuno-oncology panel (96 proteins per panel, e.g. PD-L1, IL-4, IL-12, IL-13, ng/ml).
Immunohistochemistry and Imaging Mass Cytometry/VECTRA of biopsies | from day 43 to day 155
  Biopsies will be sectioned and stained for the determination of the cutaneous homeostasis and tumor micro-environment by visualising infiltration of cellular immune subsets (e.g. presence of CD4 and CD8).
Circulating protein biomarkers by PCR amplification | from day 0 to day 155
  Blood will be drawn using a venipuncture during visits and analyzed for the presence of various chemokines and cytokines (e.g. CCL20, CCL17, CXCL8).
Cells/ml; Circulating immune cell subsets | from day 0 to day 155
  Blood will be drawn using a venipuncture during visits and analyzed for the presence of immune cells (e.g. CD4+ and CD8+ T-Cells) using flow cytometry.
Itch Tracking by Derma Track | from day 0 to day 155
  Subjects are requested to wear a smartwatch during the night to register total duration of scratch movements.
User experience and subjective burden questionnaire | from day 43 to day 155
  Measures the user experience and subjective burden of the different imaging modalities used in this study. Scores ranging from 0 (no burden) to 100 (severe burden).
Blister immune cell subsets during dermatitis reactions | from day 43 to day 155
  Blisters will be induced on the lesional skin and the blister exudate aspirated. Blister exudate will be analyzed for the presence of immune cells (e.g. CD4+ and CD8+ T-Cells) using flow cytometry.
Change from baseline in blister immune cell subsets after 16 weeks of treatment | day 43 and day 155
  Blisters will be induced on the lesional skin and the blister exudate aspirated. Blister exudate will be analyzed for the presence of immune cells (e.g. CD4+ and CD8+ T-Cells) using flow cytometry.
Blister protein biomarkers by high-throughput, multiplex immunoassays of proteins by Proximity Estension Assay (PEA) technology | from day 43 to day 155
  Blisters will be induced on the lesional skin and blister fluid aspirated. Blister fluid will be analyzed for the presence of various chemokines and cytokines using the Olink inflammation and immuno-oncology panel (96 proteins per panel, e.g. PD-L1, IL-4, IL-12, IL-13, ng/ml).
Change from baseline in blister protein biomarkers, by high-throughput, multiplex immunoassays of proteins by Proximity Estension Assay (PEA) technology | day 43 and day 155
  Blisters will be induced on the lesional skin and blister fluid aspirated. Blister fluid will be analyzed for the presence of various chemokines and cytokines using the Olink inflammation and immuno-oncology panel (96 proteins per panel, e.g. PD-L1, IL-4, IL-12, IL-13, ng/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rissmann, Prof. Dr., Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No